CLINICAL TRIAL: NCT05604105
Title: Oral Cancer Awareness Level in Egypt: a Pilot Cross-sectional Study
Brief Title: Oral Cancer Awareness in Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ayat Gamal-AbdelNaser (Other)
Collaborators: Ahram Canadian University (Other)
Responsible Party: Sponsor-Investigator, Ayat Gamal-AbdelNaser, Principle investigator, Cairo University
Organization: Cairo University (Other)
Other Study IDs: ACU-Med1
Record Dates: First submitted 2022-10-25; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sample of the Egyptian population: Participants of Giza residents.
  Inclusion criteria:
  • Adult individuals (Age>18 years).
  Exclusion criteria:
  * Dental students or dental practitioners; as awareness of the disease is an integral part of their profession.
  * Oral cancer patients: Individuals who experience currently or previously having oral cancer.
  * Individuals with mental or communication disabilities.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The questionnaire includes a section for socio-demographic data, a section to detect their general awareness of oral cancer as a disease, a section about their awareness of its signs and symptoms and lastly, a section about its risk factors and habits.

SUMMARY:
Oral cancer is a fatal disease with high prevalence and poor survival rate. Most oral cancer cases can be detected by the patients themselves. So, when a patient is aware of oral caner, the patient would realize its signs and symptom and seek early medical care; therefore, improving the prognosis.

To our knowledge, the level of awareness of oral cancer has not been investigated in Egyptian population. Therefore, this study is planned to be a pilot study as a first study in Egypt.

DETAILED DESCRIPTION:
Cancer of the oral cavity is considered a global health burden. According to GLOBOCAN report of 2012, the incidence of oral cancer in Egypt was 1,687 per 10,000 per annum; while the mortality was 659 per 10,000 per annum. Statistically, the rates are expected to increase as to reach 2,658 per 10,000 incidence and 1,069 per 10,000 mortality by the year 2030.

Fortunately, 85% of head and neck cancers are visible. Therefore, the patient does not always need to visit a specialist for a special test to check for oral cancer. Instead, if the patients have basic knowledge about oral cancer, its signs and symptoms and its risk factors, they can detect the change themselves.

As a first step to reach this amazing goal, the level of awareness of the general population needs to be detected.

To the best of our knowledge, the awareness of oral cancer has not been assessed in the general population of Egypt before. As awareness of oral cancer is mandatory for dental practitioners, our study targets the general population other than those working in the dentistry field.

ELIGIBILITY:
Inclusion criteria:

* Adult individuals (Age>18 years).

Exclusion criteria:

* Dental students or dental practitioners; as awareness of the disease is an integral part of their profession.
* Oral cancer patients: Individuals who experience currently or previously having oral cancer.
* Individuals with mental or communication disabilities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This cross-sectional study aims to quantify the awareness of Egyptian population to oral cancer. The study will be undertaken in the city of 6th of October in Giza governorate. It is a city of population 368,650 inhabitants.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Level of awareness to oral cancer | 6 months

IPD SHARING:
Plan to Share IPD: Undecided